CLINICAL TRIAL: NCT00812201
Title: Evaluation of Left Ventricular AutoThreshold
Acronym: ELEVATE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CRRT081908H
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: Heart failure; auto threshold; pacing; CRT-P or CRT-D recipients, threshold measurements
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Device: No intervention is used. Collection of signals only.

INTERVENTIONS:
Device: No intervention is used. Collection of signals only. — Device received per standard of care.

SUMMARY:
This study will collect data on a new feature for future heart failure devices via an external non-implantable system.

DETAILED DESCRIPTION:
ELEVATE is an acute, prospective, multi-center, feasibility study with a randomized within patient test sequence and pulse width, designed to characterize the performance of the Left Ventricular Auto Threshold feature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to receive a CRT-P or CRT-D, based on physician discretion
* Patients who are willing and capable of participating in all testing associated with this study
* Patients who are 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Patients who have, or are scheduled to receive a unipolar LV pace/sense lead to be used with the CRT-P/CRT-D device, unless the patient has any commercially available epicardial leads with at least two electrodes (from one or more leads)
* Patients with pre-existing leads other than those specified in this investigational plan (unless the Investigator intends to replace them with permitted leads)
* Patients with a pre-existing unipolar pacemaker that will not be explanted/abandoned
* Patients enrolled in any concurrent study, without Boston Scientific CRM written approval, that may confound the results of this study
* Patients with a prosthetic mechanical tricuspid heart valve
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to collect data to characterize the performance of the LVAT feature. | Implant

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Ellenbogen, M.D., Principal Investigator — Virginia Commonwealth University Health System
Locations (2):
- United States (2):
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Monongalia General Hospital, Morgantown, West Virginia